CLINICAL TRIAL: NCT06216756
Title: A Prospective, Open Label, Single-Arm, Multi-Center Study Evaluating Cryopreserved Osteochondral Allograft Cores for the Treatment of Osteochondral Lesions in the Knee
Brief Title: Evaluating Cryopreserved Osteochondral Allograft Cores for the Treatment of Osteochondral Lesions in the Knee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COCA-OCA-001
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Osteochondral Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteochondral transplant on the femoral condyle (Experimental): Eligible and enrolled patients will receive one or more cryopreserved osteochondral allograft core as part of their osteochondral transplant procedure
  Interventions: Procedure: osteochondral transplant on the femoral condyle

INTERVENTIONS:
Procedure: osteochondral transplant on the femoral condyle — Patients between the ages of ≥12 years and ≤ 60 years who have a symptomatic full-thickness cartilage lesion (Grade 3 or 4) on the femoral condyle, in a mechanically stable knee, or is being mechanically stabilized in the same procedure, between 0.9-8.0 cm2 in size, and cystic changes requiring osseous repair, as confirmed by MRI , CT scan, or arthroscopy and will undergo a osteochondral transplant by removing the damaged cartilage and replacing that cartilage with a cryopreserved osteochondral allograft core.

SUMMARY:
The primary objective of this study is to obtain evidence of the effectiveness of Cryopreserved Osteochondral Allograft Core in the treatment of osteochondral lesions on the femoral condyle.

DETAILED DESCRIPTION:
Patients between the ages of ≥12 years and ≤ 60 years who have a symptomatic full-thickness cartilage lesion (Grade 3 or 4) on the femoral condyle, in a mechanically stable knee, or is being mechanically stabilized in the same procedure, between 0.9-8.0 cm2 in size, and cystic changes requiring osseous repair, as confirmed by MRI , CT scan, or arthroscopy, and undergoing an osteochondral transplant procedure will be eligible for enrollment. Patients will receive one or more cryopreserved osteochondral allograft core transplants to replace damaged cartilage.

Patients will be followed for up to 60 months post-procedure (6 weeks, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months) to evaluate short and long-term outcomes of the procedure using the cryopreserved osteochondral allograft cores.

ELIGIBILITY:
Inclusion Criteria:

* Patients are ≥12 years and ≤ 60 years of age at the time of surgery.
* Symptomatic patient presenting with moderate to severe pain in the index knee - unresponsive to conservative treatment (i.e., medication, bracing, physical therapy) and/or previous surgical intervention OR unsalvageable lesion that requires transplantation at the discretion of the treating physician.
* Radiographically diagnosed, by MRI or CT scans, or through arthroscopy, to have a cartilage defect on the femoral condyle between 0.9-8.0 cm2 in size.
* Will be having an osteochondral transplant procedure.
* Has a mechanically stable knee or can be mechanically stabilized in the same procedure.
* Has a normally aligned knee as confirmed by anatomic comparison to contralateral limb, or <5° varus or valgus malalignment that has been corrected or will be corrected in same procedure.
* Ipsilateral knee compartment has intact menisci or requires partial meniscectomy ≤ 50% resulting in stable menisci.
* Confirmation MRI, CT scan, or arthroscopy obtained pre-operatively within 90 days of surgery
* Willingness to follow standardized rehabilitation procedures.
* Has the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.

Exclusion Criteria:

* Bipolar articular cartilage involvement (kissing lesions) of the ipsilateral compartment (i.e., > than ICRS Grade 2 on the opposing articular surface).
* Has had a prior osteochondral allograft transplant procedure in the same knee.
* Will be receiving a meniscus allograft transplantation in the same procedure.
* Body Mass Index (BMI)of ≥ 35 kg/m2.
* Active malignancy: undergoing treatment for tumor or boney traumatic injury or a history of any invasive malignancy (except non-melanoma skin cancer) unless the patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years.
* Clinical and/or radiographic disease in the affected joint that includes generalized osteoarthritis, gout or a history of gout or pseudo-gout.
* Active local microbial infection or a systemic infection, including HIV, syphilis, Hepatitis B or Hepatitis C.
* Currently immunologically suppressed or immunocompromised, or a medical condition requiring radiation and/or chemotherapy.
* Unstable cardiovascular, renal, hepatic, endocrine and/or pulmonary disease, cancer, or uncontrolled diabetes.
* Has a history of any inflammatory joint arthropathy.
* Currently using/chronic on oral corticosteroids.
* Received interarticular corticosteroid injection ≤ 90 days prior to surgery.
* Received hyaluronic acid injections into the joint space ≤ 45 days prior to surgery.
* Is a female patient who is pregnant.
* Physically or mentally compromised (i.e., being currently treated for a psychiatric disorder, senile dementia, Alzheimer's disease) in a manner that would compromise his/her ability to participate in the clinical study.
* Has a history of substance abuse- (including but not limited to recreational drugs, alcohol) or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an in-patient substance abuse program.
* Patients who, in the opinion of the Investigator, would not be able or willing to comply with the protocol.
* Is currently involved in a study of another investigational product for similar purpose or has been in the previous 90 days.
* Has any contraindications for MRI.
* Is having the procedure as part of a Worker's Compensation claim.
* Is a ward of the state, prisoner, or transient.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) score | 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months post procedure
  Change of physical functioning and pain from baseline as assessed by the subjective International Knee Documentation Committee (IKDC) score.
  Scores are reported on a 0-100 scale, with low scores indicating worse outcomes and higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Change from baseline (pre-operative)
  Scores are reported on a 0-100 scale, with low scores indicating worse outcomes and higher scores indicating better outcomes.
Assessment of repair cartilage structure | 12 months, 24 months and 60 months post procedure
  Assessment of repair cartilage structure, using Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scores, as measured by Magnetic Resonance Imaging (MRI).
  Scores are reported on a 0-100 scale, with low scores indicating worse outcomes and higher scores indicating better outcomes.
Graft incorporation | 12 months, 24 months and 60 months post procedure
  Assessment of graft incorporation using Magnetic Resonance Imaging (MRI)
12-item Veterans RAND (VR-12) | 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months post procedure
  Change from baseline (pre-operative)
  The instrument is primarily used to measure health related quality of life, to estimate disease burden and to evaluate disease-specific benchmarks with other populations. The 12 items are summarized into two scores, a "Physical Health Summary Measure" and a "Mental Health Summary Measure."
Revision surgery | 60 months post-procedure
  Incidences of revision surgeries during study follow up time period

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Banner- University Medical Center- Phoenix Orthopedic and Sports Medicine Institute, Phoenix, Arizona
  - Cedars-Sinai Kerlan Jobe Institute, Los Angeles, California
  - Stanford Medicine-Orthopaedics and Sports Medicine in Redwood City, Redwood City, California
  - University of California San Francisco, San Francisco, California
  - Rush Copley Medical Center, Aurora, Illinois
  - University of Kentucky Research Foundation, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No
After patients have signed the ICF and have been determined to meet the inclusion/exclusion criteria, the patient will be given a patient identification number that consists of a 2-digit site number and a 3-digit patient number. As allowed by governing privacy requirements, this will serve as a patient's identifier on all study-related documentation.